CLINICAL TRIAL: NCT00788255
Title: In-vitro Study to Assess the Coagulation Effects of Exogenous Oxytocin Using Thromboelastography.
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alex James Butwick, Principle Investigator, Stanford University
Other Study IDs: SU-10242008-1327
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Venous blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All participants: For each patient, 1 solution with citrated whole blood (control) and 3 solutions with citrated whole blood and exogenous oxytocin were prepared in separate vials using micropipettes as follows:
  Citrated whole blood 1mL + 23μU oxytocin: final exogenous oxytocin concentration=22.5 μU/mL Citrated whole blood 1mL + 31μU oxytocin: final exogenous oxytocin concentration=30.1μU/mL Citrated whole blood 1mL + 34μU oxytocin: final exogenous oxytocin concentration=32.9μU/mL
  After mixing by inversion 8-10 times, 360μL kaolin-activated blood of each study solution was pipetted into a plastic cup in a prewarmed Thromboelastograph® (37°C). Each sample was recalcified in a plastic cup with 10μL of CaCl2 6.45%, and TEG® analysis was commenced within 1 minute of reconstituted sample preparation.
  Interventions: Drug: Final exogenous oxytocin concentration=22.5 μU/mL; Drug: Final exogenous oxytocin concentration=30.1μU/mL; Drug: Final exogenous oxytocin concentration=32.9μU/mL

INTERVENTIONS:
Drug: Final exogenous oxytocin concentration=22.5 μU/mL — Citrated whole blood 1mL + 23μU oxytocin. After mixing by inversion 8-10 times, 360μL kaolin-activated blood of each study solution was pipetted into a plastic cup in a prewarmed Thromboelastograph® (37°C). Each sample was recalcified in a plastic cup with 10μL of CaCl2 6.45%, and TEG® analysis was commenced within 1 minute of reconstituted sample preparation.
  Other Names: TEG
Drug: Final exogenous oxytocin concentration=30.1μU/mL — Citrated whole blood 1mL + 31μU oxytocin. After mixing by inversion 8-10 times, 360μL kaolin-activated blood of each study solution was pipetted into a plastic cup in a prewarmed Thromboelastograph® (37°C). Each sample was recalcified in a plastic cup with 10μL of CaCl2 6.45%, and TEG® analysis was commenced within 1 minute of reconstituted sample preparation.
  Other Names: TEG
Drug: Final exogenous oxytocin concentration=32.9μU/mL — Citrated whole blood 1mL + 34μU oxytocin. After mixing by inversion 8-10 times, 360μL kaolin-activated blood of each study solution was pipetted into a plastic cup in a prewarmed Thromboelastograph® (37°C). Each sample was recalcified in a plastic cup with 10μL of CaCl2 6.45%, and TEG® analysis was commenced within 1 minute of reconstituted sample preparation.
  Other Names: TEG

SUMMARY:
Oxytocin is normally administered following delivery in pregnant patients to reduce postpartum bleeding by increasing uterine tone. It is unclear whether the use of intravenous oxytocin alters coagulation in pregnant patients. The purpose of the in-vitro study is to assess the coagulation changes of oxytocin in blood samples from pregnant patients using thromboelastrography (TEG). TEG is a point-of-care device which measures the viscoelastic properties of clot formation, and can provide rapid and detailed information about coagulation changes. We aim to collect blood samples from pregnant patients to assess the in-vitro effects of synthetic oxytocin on coagulation using TEG.

DETAILED DESCRIPTION:
All obstetric patients presenting for elective induction of labor or elective Cesarean delivery will be informed about the study prior to and on admission to the labor and delivery unit. Admission blood sampling will take place by venepuncture for the following analysis:TEG, PT, PTT, INR, Hct, Platelet count.The results of oxytocin influence on thromboelastogram parameters will be compared to a control. The control is an aliquot of parturient blood with no added oxytocin. Thromboelastography will be used to assess coagulation changes between control samples and blood samples with added oxytocin. The results will not be used to influence clinical management of any case.

ELIGIBILITY:
Inclusion Criteria:All obstetric patients with singleton pregnancies admitted to the labor and delivery unit at Lucile Packard Childrens Hospital awaiting elective induction of labor or elective Cesarean delivery. We will select 25 healthy ASA 1 patients with singleton pregnancies who are scheduled for uncomplicated elective induction of labor. Gestational age equal to or greater than 37 weeks.

Exclusion Criteria:Patients with underlying coagulation disorders. Patients with thrombocytopenia. Patients with pregnancy-induced hypertension, pre-eclampsia. Patients admitted for non-elective cesarean section. Patients in active labor. Patients requiring the following medications prior to surgery: NSAIDS, aspirin, anticoagulants.

Patients with significant obstetric or medical disease. No patients <18 years of age will be recruited.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: healthy pregnant patients awaiting elective induction of labor or cesarean delivery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Butwick, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 25
Oxytocin Infusion 1: 22.5 μU/mL | 25
Oxytocin Infusion 2: 30.1μU/mL | 25
Oxytocin Infusion 3: 32.9μU/mL | 25
Oxytocin: 0 μU/mL | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All blood samples for this study were taken from a total cohort of 25 patients
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Our cohort comprised healthy adult pregnant women
  Participants
    <=18 years | 0
    Between 18 and 65 years | 25
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: r Time
Description: thromboelastographic indices - reaction time (normal range, 5-10 min)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | All Participants
Number analyzed (Participants) | 25
minutes
  Exogenous Oxytocin 22.5 | 5.6 (1.4)
  Exogenous Oxytocin 30.1 | 4.2 (1.3)
  Exogenous Oxytocin 32.9 | 3.9 (1.3)
  Exogenous oxytocin 0 | 6 (1.5)

2. Primary Outcome: k Time
Description: thromboelastographic indices - clot formation time (normal range, 1-3 min)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | All Participants
Number analyzed (Participants) | 25
minutes
  Exogenous Oxytocin 22.5 | 1.6 (0.4)
  Exogenous Oxytocin 30.1 | 1.5 (0.7)
  Exogenous Oxytocin 32.9 | 1.4 (0.4)
  Exogenous Oxytocin 0 | 1.7 (0.4)

3. Primary Outcome: Alpha Angle
Description: thromboelastographic - alpha angle = clot formation rate (normal range, 53 degress to 72 degrees)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | All Participants
Number analyzed (Participants) | 25
degrees
  Exogenous Oxytocin 22.5 | 67.4 (4.2)
  Exogenous Oxytocin 30.1 | 67.7 (3.7)
  Exogenous Oxytocin 32.9 | 69.4 (4.2)
  Exogeneous oxytocin 0 | 66.2 (4.4)

4. Primary Outcome: MA
Description: thromboelastographic indices - maximum amplitude (normal range, 50-70 mm)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 25
mm
  Exogenous Oxytocin 22.5 | 69.8 (4.3)
  Exogenous Oxytocin 30.1 | 67.2 (3.7)
  Exogenous Oxytocin 32.9 | 69.0 (4.2)
  Exogeneous Oxytocin 0 | 67.2 (3.9)

5. Primary Outcome: MRTG
Description: thromboelastographic indices - maximum rate of thrombus generation (normal range, 5-17 mm/min)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm/min
Arm/Group | All Participants
Number analyzed (Participants) | 25
mm/min
  Exogenous Oxytocin 22.5 | 13.5 (2.7)
  Exogenous Oxytocin 30.1 | 14.9 (3.7)
  Exogenous Oxytocin 32.9 | 14.3 (2.8)
  Exogeneous Oxytocin 0 | 12.8 (2.5)

6. Primary Outcome: Tmax
Description: thromboelastographic indices - time to initiation of clot formation plus time to achieve maximum rate of clot strength development (normal range, 6-12 min)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | All Participants
Number analyzed (Participants) | 25
minutes
  Exogenous Oxytocin 22.5 | 6.9 (1.6)
  Exogenous Oxytocin 30.1 | 5.4 (1.9)
  Exogenous Oxytocin 32.9 | 5.0 (1.5)
  Exogeneous Oxytocin 0 | 7.5 (1.7)

7. Primary Outcome: TTG
Description: thromboelastographic indices - total thrombus generation (normal range, 584-796 mm)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Participants
Number analyzed (Participants) | 25
mm
  Exogenous Oxytocin 22.5 | 845.9 (53.9)
  Exogenous Oxytocin 30.1 | 820 (45.9)
  Exogenous Oxytocin 32.9 | 839.7 (51.8)
  Exogeneous Oxytocin 0 | 819.4 (48.9)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- 22.5 μU/mL Exogenous Oxytocin; 30.1 μU/mL Exogenous Oxytocin; 32.9 μU/mL Exogenous Oxytocin: thromboelastography: TEG was performed on kaolin-activated citrated blood samples
- 0 μU/mL Exogenous Oxytocin: Thromboelastography on native blood sample.
Arm/Group | 22.5 μU/mL Exogenous Oxytocin | 30.1 μU/mL Exogenous Oxytocin | 32.9 μU/mL Exogenous Oxytocin | 0 μU/mL Exogenous Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No